CLINICAL TRIAL: NCT04165252
Title: Evaluation of the Relationship Between Vaginal, Placental and Neonatal Mycobiota and Microbiome With Preterm Birth in Women With Short Cervical Length
Brief Title: Vaginal, Placental and Neonatal Buccal Mycobiota and Microbiome in Preterm Birth
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Koç University (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Sponsor
Other Study IDs: 119S463
Record Dates: First submitted 2019-10-14; First posted 2019-11-15 (Actual); Last update posted 2021-06-02 (Actual); Status verified 2021-03

CONDITIONS: Preterm Birth; Microbial Colonization
Keywords: Preterm birth; Microbiota; Mycobiota; Short Cervix; Progesterone
MeSH Terms: conditions — Premature Birth; Communicable Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 41 Weeks
Biospecimen Retention: Samples With DNA — Maternal (vaginal), neonatal (buccal) and placental specimens will be collected. Genomic DNA will be stored at -80 ℃ until the analysis of microbiota and mycobiota are performed by using BIO PowerSoil DNA isolation kits.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Term Birth: Delivery between 37-41 weeks of gestation
  Interventions: Diagnostic Test: Collection of vaginal, neonatal buccal and placental samples
- Preterm birth: Delivery between 24-37 weeks of gestation
  Interventions: Diagnostic Test: Collection of vaginal, neonatal buccal and placental samples

INTERVENTIONS:
Diagnostic Test: Collection of vaginal, neonatal buccal and placental samples — Analysis of microbiome and mycobiota of vaginal, neonatal buccal and placental

SUMMARY:
Microbiota contributes to the immunological, hormonal and metabolic homeostasis of the host. As in all natural orifices in the body, there is also a microbiota and mycobiota specific to the vagina.

On the other hand, the sonographic short cervix in the second trimester of pregnancy is associated with preterm delivery, which may be an important cause of mortality and morbidity in the neonatal period. American Society of Obstetricians and Gynecologists (ACOG), British Royal Society of Obstetricians and Gynecologists (RCOG) and the American Society of Maternal Fetal Medicine (SMFM) suggest that the measurement of transvaginal sonographic cervical length at 20-24 gestational weeks for the screening of preterm birth. The aforementioned associations also recommend the use of progesterone in the treatment of women who diagnosed with short cervix by transvaginal ultrasonography due to the fact that progesterone is an effective medication in the prevention of preterm birth (Grade B).

Previous vaginal microbiota studies have shown that some bacterial species such as Lactobacillus insers cause a predisposition to premature labor in women with a short cervix. However, the prominent lack in these studies is that the eukaryotic fungi in abundant vaginal flora have not been evaluated.

On the other hand, it was already shown that progesterone treatment is able to prevent only 45% preterm birth in women with short cervical length. This observational prospective study thus aims to evaluate the variety of microbiota and/or mycobiota in pregnancies resulting in preterm birth and those who give birth at term. Although women with short cervical length receive progesterone regularly from the second trimester, the preterm birth may occur. In this study, the investigators also aim to evaluate the patterns of microbiota and mycobiota from vaginal swabs of women who had preterm birth with short cervical length and postpartum swabs of the placenta and fetal oral cavity.

DETAILED DESCRIPTION:
Preterm birth is responsible for more than 70% of all neonatal and infant deaths. In addition, the risk of cerebral palsy among children born preterm is 10 times than those born at term. The risk of preterm birth is inversely related to cervical length at midgestation. Randomized-controlled trials involving singleton pregnancies with a short cervical length ( less than 25 mm) have shown that the prophylactic use of progesterone significantly decrease the rate of preterm delivery and neonatal death. The relation of vaginal micobiota with preterm birth has been documented. Yet, impact of short cervical lenght and progesteron treatment on vaginal, neonatal and placental microbiota and mycobiota has not been evaluated. The objectives of present study are to adress the following points;

1. Longitudinal maternal (vaginal), fetal (oral) and placental (basal plate and parenchyma) 16S-based and 18S-based metagenomic profiling with inferred metagenomics will reveal distinct microbial communities in association with preterm birth.
2. Comparison of vaginal, neonatal (buccal) and placental (basal plate and parenchyma) 16s rRNA with bacteria and 18s rRNA with fungi in pregnant women with a short cervical length with those with normal cervical length;

2. Comparison of maternal (vaginal), neonatal(oral) and placental (basal plate and parenchyma)16s rRNA with bacteria and 18s rRNA with fungi in pregnant women with short cervical length who gave a preterm birth with those who gave birth at term; 3. The effect of progesterone on maternal (vaginal), neonatal (buccal) and placental (basal plate and parenchyma)16s rRNA with bacteria and 18s rRNA with fungi.

The measurements of cervical length will be performed in two different periods of pregnancy (11-14 and 18-22 weeks of gestation) in singleton pregnancies. Firstly, the vaginal swabs will be collected from women who accept to participate in the study at 11-14th weeks of gestation just before the measurement of cervical length. Also, the vaginal swabs will be done again at 18-22 weeks of gestation as explained above. Micronized progesterone will be started in women with a cervical length equal or less than 25 mm (smaller than 3rd percentile) at 18-22 weeks of gestation. The medication (progesterone 200mg) will be administered intravaginally every night before bedtime and will continue until 36th gestational week unless the patient gives birth. Measurement of cervical length will be repeated transvaginally at 28th and 32nd gestational weeks, and samples will be obtained with a cervical swab before these measurements. In order to evaluate the presence of placental mycobiota and microbiota, 1 cm x 1 cm x 1 cm of the tissue sample from the placenta that is 3 cm lateral of the cord insertion will be taken under sterile conditions after birth. In order to evaluate the amniotic compartment, a buccal mucosal swab will be collected from the neonates immediately after birth. All samples will be delivered to our Research Laboratory immediately and stored in -80 ℃ cabinet until the evaluation. The V3-V4 regions by the 16s ribosomal RNA sequencing method will be sequenced with the Illumina MiSeq device and the data will be analyzed according to the protocols standardized in the Human Microbiome Project.

DNA samples that will be ranked from the data to be sequenced in accordance with the ITS1 region metabiota protocol will be evaluated within the Human Microbiome Project.

Pseudomonas, Escherichia, Neisseria, Streptococcus, Lactobacillus, Candida, Actinomyces will be used as positive controls and, V3-V4 and ITS regions will be matched for bacterial microbiota and Fungal microbiota. After the "Operational taxonomic units" of the amplicons are configured with the VSEARCH program, the analyzes will be carried out with GENBANK microbiota and micobiota data.

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnancies
* The subject has voluntarily signed the Informed Consent Form and associated forms after having the contents explained

Exclusion Criteria:

* Multiple pregnancies
* The presence of a major fetal anomaly or known chromosomal abnormality
* Finding the intrauterine mort de fetus
* Antibiotic and/or antifungal use within two weeks at the collection of samples
* Pregnant women under 18 years of age
* Women with previous cervical surgery
* Women who do not accept to participate to be in the study
* The presence of a uterine anomaly
* Women with vaginal bleeding at the time of cervical swabs taken

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Pregnant women attending prenatal clinics of Koc University Hospital in Istanbul.
Sampling Method: Probability Sample
Enrollment: 92 (Estimated)
Dates: Start 2020-04-01 (Actual); Primary Completion 2021-12-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Characterization of Maternal-Fetal microbiome and mycobiome | 11 weeks of gestation to date of delivery
  Characterize the maternal(vaginal), placental, and neonatal (buccal) microbiome and mycobiome in a cohort at risk of preterm birth by using the BIO Power Soil DNA Isolation kit. The investigators will able to evaluate whether there is an association between microbiome and mycobiome changes with preterm birth. The V3-V4 regions by the 16s rRNA and ITS regions by 18s rRNA sequencing method will be sequenced. After the "Operational taxonomic units" of the amplicons are configured with the VSEARCH program, the analyzes will be carried out with GENBANK microbiota and micobiota data.

SECONDARY OUTCOMES:
The effect of progesterone on maternal microbiome (vaginal and placenta) with progesterone | 11 weeks of gestation to date of delivery
  Characterize the maternal, placental, and neonatal microbiome in a cohort at risk of preterm birth who receive progesterone treatment. Not all the women will ultimately deliver at term despite of prophylactic management of progesterone; the investigators will be able to see if there are microbiome changes associated with preterm birth by using the BIO Power Soil DNA Isolation kit. We will able to evaluate whether there is an association between microbiome and mycobiome changes with preterm birth. The V3-V4 regions by the 16s rRNA and ITS regions by 18s rRNA sequencing method will be sequenced. After the "Operational taxonomic units" of the amplicons are configured with the VSEARCH program, the analyzes will be carried out with GENBANK microbiota and micobiota data.
Variety of microbial and mycobial fingerprintings | 11 weeks of gestation to date of delivery
  Comparison of vaginal, neonatal buccal and placental 16S rRNA and 18S rRNA gene sequencing between women with a short cervix who give a preterm birth with those who deliver at term.

CONTACTS AND LOCATIONS:
Overall Officials: Ebru Celik, M.D., Study Director — Koç University; Fusun Can, M.D., Study Director — Koc University School of Medicine; Mert Turgal, M.D., Principal Investigator — Koc University School of Medicine; Ozlem Dogan, M.D., Principal Investigator — Koc University School of Medicine; Mehmet Gonen, P.h.D, Principal Investigator — Koc University School of Medicine; Tugba Gursoy, M.D., Principal Investigator — Koc University School of Medicine
Locations (1):
- Koc University Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
The recruitment of participants will begin on November 2019 and the anticipated date for the completion of the study is November 2022.
Supporting Information: Study Protocol, ICF, CSR, Analytic Code
Time Frame: The data will be available for 5 years
Access Criteria: The researchers who are responsible for the recruitment of patients will have access code. The web address will be ready in November 2019 and the researcher will have a personal ID and password to enter the participants' data.

REFERENCES:
- [Background] Aagaard K, Ma J, Antony KM, Ganu R, Petrosino J, Versalovic J. The placenta harbors a unique microbiome. Sci Transl Med. 2014 May 21;6(237):237ra65. doi: 10.1126/scitranslmed.3008599. PMID 24848255
- [Background] DiGiulio DB, Romero R, Amogan HP, Kusanovic JP, Bik EM, Gotsch F, Kim CJ, Erez O, Edwin S, Relman DA. Microbial prevalence, diversity and abundance in amniotic fluid during preterm labor: a molecular and culture-based investigation. PLoS One. 2008 Aug 26;3(8):e3056. doi: 10.1371/journal.pone.0003056. PMID 18725970
- [Background] Gardella C, Riley DE, Hitti J, Agnew K, Krieger JN, Eschenbach D. Identification and sequencing of bacterial rDNAs in culture-negative amniotic fluid from women in premature labor. Am J Perinatol. 2004 Aug;21(6):319-23. doi: 10.1055/s-2004-831884. PMID 15311367
- [Background] Han YW, Shen T, Chung P, Buhimschi IA, Buhimschi CS. Uncultivated bacteria as etiologic agents of intra-amniotic inflammation leading to preterm birth. J Clin Microbiol. 2009 Jan;47(1):38-47. doi: 10.1128/JCM.01206-08. Epub 2008 Oct 29. PMID 18971361
- [Background] Iams JD, Goldenberg RL, Meis PJ, Mercer BM, Moawad A, Das A, Thom E, McNellis D, Copper RL, Johnson F, Roberts JM. The length of the cervix and the risk of spontaneous premature delivery. National Institute of Child Health and Human Development Maternal Fetal Medicine Unit Network. N Engl J Med. 1996 Feb 29;334(9):567-72. doi: 10.1056/NEJM199602293340904. PMID 8569824
- [Background] Kindinger LM, Bennett PR, Lee YS, Marchesi JR, Smith A, Cacciatore S, Holmes E, Nicholson JK, Teoh TG, MacIntyre DA. The interaction between vaginal microbiota, cervical length, and vaginal progesterone treatment for preterm birth risk. Microbiome. 2017 Jan 19;5(1):6. doi: 10.1186/s40168-016-0223-9. PMID 28103952
- [Background] Society for Maternal-Fetal Medicine (SMFM). Electronic address: pubs@smfm.org; McIntosh J, Feltovich H, Berghella V, Manuck T. The role of routine cervical length screening in selected high- and low-risk women for preterm birth prevention. Am J Obstet Gynecol. 2016 Sep;215(3):B2-7. doi: 10.1016/j.ajog.2016.04.027. Epub 2016 Apr 28. PMID 27133011
- [Background] American College of Obstetricians and Gynecologists' Committee on Practice Bulletins-Obstetrics. Practice Bulletin No. 171: Management of Preterm Labor. Obstet Gynecol. 2016 Oct;128(4):e155-64. doi: 10.1097/AOG.0000000000001711. PMID 27661654
- [Background] Romero R, Nicolaides KH, Conde-Agudelo A, O'Brien JM, Cetingoz E, Da Fonseca E, Creasy GW, Hassan SS. Vaginal progesterone decreases preterm birth </= 34 weeks of gestation in women with a singleton pregnancy and a short cervix: an updated meta-analysis including data from the OPPTIMUM study. Ultrasound Obstet Gynecol. 2016 Sep;48(3):308-17. doi: 10.1002/uog.15953. Epub 2016 Jul 19. PMID 27444208
- [Result] DiGiulio DB, Romero R, Kusanovic JP, Gomez R, Kim CJ, Seok KS, Gotsch F, Mazaki-Tovi S, Vaisbuch E, Sanders K, Bik EM, Chaiworapongsa T, Oyarzun E, Relman DA. Prevalence and diversity of microbes in the amniotic fluid, the fetal inflammatory response, and pregnancy outcome in women with preterm pre-labor rupture of membranes. Am J Reprod Immunol. 2010 Jul 1;64(1):38-57. doi: 10.1111/j.1600-0897.2010.00830.x. Epub 2010 Mar 21. PMID 20331587

DOCUMENTS (1):
  • Study Protocol (2019-03-01): https://cdn.clinicaltrials.gov/large-docs/52/NCT04165252/Prot_000.pdf